CLINICAL TRIAL: NCT02705859
Title: Phase Ib/II Clinical Trial of Copanlisib in Combination With Trastuzumab in Pretreated Recurrent or Metastatic HER2-positive Breast Cancer
Brief Title: Phase Ib/II Trial of coPANlisib in Combination With Trastuzumab in HER2-positive Breast Cancer. (Panther Study)
Acronym: Panther
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICORG 15-02
Record Dates: First submitted 2016-02-11; First posted 2016-03-11 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: HER2 Positive Breast Cancer
MeSH Terms: interventions — copanlisib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): This study is a Phase Ib/II open label, single arm, adaptive multi-centre trial.
  Patients with HER2-positive, metastatic or incurable recurrent breast cancer, following disease progression during, or after, treatment with at least one systemic treatment regimen in the metastatic or recurrent setting, will be treated with copanlisib (at 30, 45 or 60 mg flat dosing IV weekly - depending on the maximum tolerated dose (MTD) determined in the Phase Ib part of the study) plus trastuzumab (4 mg/kg IV Cycle 1 Day 1 and then 2 mg/kg IV weekly starting from day 8).
  Interventions: Drug: Copanlisib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Copanlisib — Copanlisib is supplied as lyophilized preparation in a 6mL injection vial. The total amount of copanlisib per vial is 60mg. The solution for IV infusions is obtained after reconstitution with normal saline solution. Copanlisib will be administered on Days 1, 8 and 15 of each 28-day cycle. Copanlisib will be administered first over 60 minutes followed by the infusion of trastuzumab.
  Other Names: BAY80-6946
Drug: Trastuzumab — Trastuzumab IV weekly (4mg/kg on Cycle 1 Day 1 followed by 2 mg/kg IV weekly from Day 8).
  Other Names: Herceptin

SUMMARY:
This study is a Phase Ib/II open label, single arm, adaptive multi-centre trial of copanlisib in combination with trastuzumab in pretreated recurrent or metastatic HER2-positive breast cancer.

Patients with HER2 positive, metastatic or incurable recurrent breast cancer, following disease progression during, or after, treatment with at least one systemic treatment regimen in the metastatic or recurrent setting, will be treated with copanlisib (at 30, 45 or 60 mg flat dosing IV weekly - depending on the maximum tolerated dose (MTD) determined in the Phase Ib part of the study) plus trastuzumab (4 mg/kg IV Cycle 1 Day 1 and then 2 mg/kg IV weekly starting from day 8).

DETAILED DESCRIPTION:
Phase Ib One of three dose levels of copanlisib is assigned at registration according to the dose escalation scheme.

Phase II The copanlisib dose for the Phase II part of the trial will be based on the MTD established in the Phase Ib part of the study.

Clinical and laboratory parameters will be assessed to evaluate disease response and toxicity of study therapy.

Safety assessments will be performed throughout the study.

Efficacy assessments (radiological examination) will be performed on all patients every 8 weeks for the first 24 weeks and every 12 weeks thereafter.

Following baseline cardiac assessment, cardiac safety monitoring will include physical exam (with New York Heart Association (NYHA) functional classification for patients with diagnosed congestive heart failure) during each cycle, Multigated acquisition (MUGA) scan or Echocardiogram (ECHO) and 12 lead Electrocardiogram (ECG) within 7 days of Day 1 of every third cycle starting at cycle 3 (Cycle 3, Cycle 6, etc.).

ELIGIBILITY:
Inclusion Criteria

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Adult women ≥ 18 years of age.
2. Histologically confirmed HER2-positive breast cancer:

   Documented HER2 overexpression by local laboratory (IHC 3+ or FISH or CISH positive).

   IHC 3+ or FISH/CISH positive on diagnostic breast biopsy or surgical breast resection sample or metastatic disease site biopsy.
3. Recurrent incurable or metastatic breast cancer:

   Eligible recurrent disease is recurrent disease that is considered incurable by the treating oncologist. Many local-only recurrences are treated with curative intent; a treatment plan with curative intent for a local-only recurrence would indicate that the patient is not eligible for this clinical trial. A local-only recurrence must be considered incurable by the treating oncologist for the patient to be eligible.
4. At least one measurable lesion according to RECIST criteria (Version 1.1). Patients with bone only disease are not eligible.
5. Patient has received at least one trastuzumab-based or T-DM1-based treatment regimen in the setting of metastatic disease or incurable locoregional recurrence. A trastuzumab-based or T-DM1-based treatment regimen is considered as any treatment regimen that includes trastuzumab or T-DM1.

   Patients must have had at least 1 line of therapy for metastatic and/or incurable locoregional recurrent disease to be eligible. A patient is eligible regardless of the period of time from adjuvant therapy so long as she has disease that is progressing after at least 1 line of trastuzumab-based therapy in the setting of metastatic disease and/or incurable locoregional recurrence.
6. Disease progression during or following at least 1 prior trastuzumab-based or trastuzumab emtansine (T-DM1) based treatment regimen in the setting of metastatic disease or incurable locoregional recurrence.
7. ECOG performance status ≤ 2.
8. Life expectancy of at least 3 months.
9. Availability of fresh tissue and/or archival tumour tissue at screening.
10. Women of childbearing potential must agree to use a highly effective method of contraception when sexually active. This applies from signing of the informed consent form until at least 100 days after the last study drug administration. The investigator or a designated associate is required to advise the patient how to achieve an adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

    i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

    ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable).

    iii. Intrauterine device (IUD).

    iv. Intrauterine hormone-releasing system (IUS).

    v. Bilateral tubal occlusion.

    vi. Successfully vasectomised partner.

    vii. Sexual abstinence.
11. Adequate baseline laboratory values collected no more than 14 days before starting study treatment:

    Total bilirubin ≤ 1.5 x ULN (< 3 x ULN for patients with metastatic disease in the liver).

    Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN (≤ 5 x ULN for patients with liver involvement from breast cancer).

    Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, this evaluation may be repeated once after at least 24 hours either according to the MDRD abbreviated formula or by 24 hour sampling. If the later result is within acceptable range, it may be used to fulfil the inclusion criteria instead.

    International normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1.5 x ULN. Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior underlying coagulopathy disorder. Close monitoring of these patients (Day 15 of Cycle 1 and Day 1 of each cycle) will be performed until INR/PTT is stable based on a measurement that is pre- dose as defined by the local standard of care.

    Platelet count ≥ 75 x 109/L. For patients with breast cancer bone marrow infiltration, platelet count ≥ 50 x 109/L.

    Haemoglobin (Hb) ≥ 8 g/dL.

    Absolute neutrophil count (ANC) ≥ 1 x 109/L. For patients with malignant bone marrow infiltration, ANC count ≥ 0.75 x 109/L.

    Fasting blood glucose ≤ 6.0 mmol/L if not diabetic or ≤ 8.9 mmol/L if diabetic.
12. Left ventricular ejection fraction (LVEF), at or above the Institutions lower limit of normal, as determined by ECHO or MUGA.
13. Patients must have recovered from clinically significant side effects associated with prior radiotherapy and chemotherapy with the exception of fatigue or neuropathy.

Exclusion criteria

Patients who meet any of the following criteria at the time of screening will be excluded from study registration:

1. Known breast cancer involvement of the brain, unless adequately controlled based on the clinical judgement of the treating physician.
2. Congestive heart failure > New York Heart Association (NYHA) class II.
3. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before registration.
4. Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion).
5. Uncontrolled Type I or II diabetes mellitus. Defined as HbA1c > 8.5% as determined during screening laboratory assessments.
6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before registration.
7. Non-healing wound, ulcer, or bone fracture.
8. Active, clinically serious infections > CTCAE Grade 2 (CTCAE v4.0).
9. Known history of human immunodeficiency virus (HIV) infection.
10. Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratory panel. Patients who test positive for Hepatitis B surface Antigen (HBsAg) or Hepatitis B core Antibody (HBcAb) will be eligible if they are negative for HBV-DNA; patients who test positive for anti-HCV antibody will be eligible if they are negative for HCV- RNA.
11. Patients with CMV PCR positive.
12. Patients with seizure disorder requiring medication.
13. Patients with evidence or history of bleeding diathesis. Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study treatment.
14. Proteinuria of Grade 3 or higher (CTCAE v4.0). Patient will be excluded if > 2+ on urinalysis (unless 24hr collection shows 24 hour urinary protein < 3.5g/24hrs).
15. History or concurrent condition of interstitial lung disease of any severity, and/or severely impaired lung function (as judged by the investigator).
16. Concurrent diagnosis of pheochromocytoma.
17. Pregnant or breast-feeding patients. Women of childbearing potential must have a serum or urine pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
18. Unresolved toxicity higher than CTCAE Grade 1 attributed to any prior therapy/procedure, excluding alopecia, peripheral neuropathy, and bone marrow parameters.
19. Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation.
20. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
21. Any illness or medical conditions that are unstable or could jeopardize the safety of patients and their compliance in the study.
22. Patients permanently withdrawn from study participation will not be allowed to re- enter the study.

    Excluded previous therapies and medications:
23. Treatment with investigational drugs other than PI3K inhibitors less than 28 days before start of treatment.
24. Ongoing immunosuppressive therapy.
25. Radiotherapy or immuno-/chemotherapy less than 4 weeks (28 days) before start of treatment.
26. Myeloid growth factors less than 7 days before start of treatment.
27. Blood or platelet transfusion less than 7 days before start of treatment.
28. Ongoing systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent. Previous corticosteroid therapy must be stopped or reduced to the allowed dose 7 days before performing the screening CT scan (or PET-CT/MRI as per RECIST 1.1) and again prior to the first study drug administration. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the minimum allowed dose before the screening. Patients may continue to use topical or inhaled corticosteroids.
29. History of having received an allogeneic bone marrow or organ transplant.
30. Major surgical procedure or significant traumatic injury (as judged by the investigator) less than 28 days before start of treatment. This does not include the study-specific biopsy.
31. Anti-arrhythmic therapy (beta blockers or digoxin are permitted).
32. Use of strong inhibitors of CYP3A4 is prohibited from Day -14 of Cycle 1 until the Safety follow up visit.
33. Use of inducers of CYP3A4 is prohibited from Day -14 of Cycle 1 until the Safety follow up visit.

Zoledronate or denosumab for patients with bone metastasis is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04; Primary Completion 2021-05 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of copanlisib in combination with trastuzumab measured by the incidence of dose limiting toxicity (DLT) of copanlisib in combination with trastuzumab within the 1st cycle at each dose level. | 1 year
Clinical Benefit Rate, defined as complete response (CR) or partial response (PR) at any time-point on the study; or stable disease (SD) lasting at least 24 weeks based on radiological assessment. | 1 year

SECONDARY OUTCOMES:
Incidences of adverse events and toxicities. | 1.5 - 2 year
Overall survival | 1.5 -2 year
Progression-Free Survival (PFS) assessed according to RECIST criteria version 1.1 | 1.5-2 year
Time to Treatment Failure (TTF) is defined as time from registration to discontinuation of therapy or add-on of new anti-cancer therapy for any reason (including death, progression and toxicity). | 1.5-2 year
Confirmed tumour response rate as assessed by RECIST criteria version 1.1. | 1.5-2 year
Duration of response (DR) as assessed by RECIST criteria version 1.1. | 1.5-2 year
To evaluate the safety and tolerability of this regimen as measured by incidence of adverse events reported and toxicity evaluation as per the NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0). | 1.5-2 year
To assess the incidence of cardiotoxicity. Cardiac safety monitoring will include physical exam, (with NYHA functional classification for patients with diagnosed congestive heart failure) at each cycle, and MUGA scan or ECHO | 1.5-2 year

CONTACTS AND LOCATIONS:
Overall Officials: Cancer Trials Ireland Dublin 11, Ireland, Study Director — Cancer Trials Ireland
Locations (3):
- Ireland (3):
  - Cancer Trials Ireland Investigative Site, Cork
  - Cancer Trials Ireland Investigative Site, Dublin
  - Cancer Trials Ireland Investigative Site, Galway

IPD SHARING:
Plan to Share IPD: Undecided